CLINICAL TRIAL: NCT02516748
Title: Prospective Study of Real-time Diagnosis of Colorectal Polyps Using Narrow-Band Imaging: Gangnam-ReaDi Study
Brief Title: Real-time Diagnosis of Colorectal Polyps Using Narrow-Band Imaging
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Su Jin Chung, Associated Professor, Seoul National University Hospital
Other Study IDs: H-1505-019-670
Record Dates: First submitted 2015-07-30; First posted 2015-08-06 (Estimated); Last update posted 2017-12-15 (Actual); Status verified 2017-12

CONDITIONS: Colon Polyps
Keywords: optical diagnosis; narrow band image
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Feedback — Less experienced endoscopists in optical diagnosis will receive feedbacks about their own accuracy of optical diagnosis.
  Other Names: Behavior change intervention

SUMMARY:
Accurate optical diagnosis of colorectal polyps could allow a "resect and discard" strategy with surveillance intervals determined based on the results of the optical biopsy. The investigators perform education to characterize the histology of diminutive and small colorectal polyps by using narrow band imaging (NBI). After education program, the investigators prospectively evaluate real-time optical biopsy analysis of polyps with NBI by 15 gastroenterologists at a medical check up center.

DETAILED DESCRIPTION:
This study is an extension of quality assurance program in Seoul National University Hospital Healthcare System Gangnam Center. This study is composed of four periods.

First, a computer based education program on the accuracy of predicting polyp histology with NBI (NICE and WASP classification) will be performed by 15 endoscopists (less experienced in NBI) during Septepber 2015.

In the second period from October 2015 till Deceber 2015, 1st phase real- time optical diagnosis for diminutive and small colorectal polyps will be activated. All endoscopists will have weekly feedback on their accuracy of optical diagnosis for polyps, and discuss the NBI findings that mismatched by histologic diagnosis all together per one month.

Third, the result of 1st phase real-time optical diagnosis will be analyzed from January 2016 till April 2016. In this period, endoscopists with low accuracy of 1st phase real-time optical diagnosis will be re-educated.

The last period from May 2016 till September 2016, 2nd phase real-time optical diagnosis for polyps will be activated. Performance will be evaluated by comparing optically predicted diagnosis with actual histologic diagnosis. Cumulative sum analysis will be used to determine the learning curve for each endoscopist. Negative predictive value for the prediction of nonneoplastic polyp and concordance of surveillance intervals for diminutive polyps diagnosed optically with high confidence will also be measured.

ELIGIBILITY:
Inclusion Criteria:

* Customers who received screening and surveillance colonoscopy in Seoul National University Hospital Healthcare System Gangnam Center from October 2015 to September 2016.

Exclusion Criteria:

* Age <18 years
* Customers who refused to offer their health check up data
* History of inflammatory bowel disease
* History of familial adenomatous polyposis
* Customers who received Incomplete colonoscopy
* History of previous colorectal resection
* Incomplete data collection on optical diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Customers who received colonoscopy for screening and surveillance of colorectal neoplasia in Seoul National University Hospital Healthcare System Gangnam Center from October 2015 to September 2016.
Sampling Method: Non-Probability Sample
Enrollment: 3268 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Concordance rate between optical diagnosis and histologic diagnosis for polyps <10 mm in real-time colonoscopy | 12 month

SECONDARY OUTCOMES:
Concordance rate in surveillance intervals of follow-up colonoscopy between optical diagnosis and histological diagnosis for polyps assessed with high confidence | 12 months
Negative predictive value for neoplastic polyps in rectosigmoid polyps 5mm or smaller with assessed high confidence | 12 months
  Negative predictive value for neoplastic polyps defined as: number of hyperplastic polyps assessed by histologic diagnosis / number of hyperplastic polyps assessed by optical diagnosis
The learning curve of accuracy of optical diagnosis | 12 months
The maintance of accuracy of optical diagnosis | 12 months
Adenoma detection rate | 24 month
Serrated lesion detection rate | 24 month

CONTACTS AND LOCATIONS:
Overall Officials: Su Jin Chung, M.D., Ph.D., Principal Investigator — Department of Internal Medicine and Healthcare Research, Healthcare System, Seoul National University Hospital
Locations (1):
- Healthcare System Gangnam Center, Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] McGill SK, Evangelou E, Ioannidis JP, Soetikno RM, Kaltenbach T. Narrow band imaging to differentiate neoplastic and non-neoplastic colorectal polyps in real time: a meta-analysis of diagnostic operating characteristics. Gut. 2013 Dec;62(12):1704-13. doi: 10.1136/gutjnl-2012-303965. Epub 2013 Jan 7. PMID 23300139
- [Background] Hassan C, Pickhardt PJ, Rex DK. A resect and discard strategy would improve cost-effectiveness of colorectal cancer screening. Clin Gastroenterol Hepatol. 2010 Oct;8(10):865-9, 869.e1-3. doi: 10.1016/j.cgh.2010.05.018. Epub 2010 Jun 1. PMID 20621680
- [Background] Ignjatovic A, East JE, Suzuki N, Vance M, Guenther T, Saunders BP. Optical diagnosis of small colorectal polyps at routine colonoscopy (Detect InSpect ChAracterise Resect and Discard; DISCARD trial): a prospective cohort study. Lancet Oncol. 2009 Dec;10(12):1171-8. doi: 10.1016/S1470-2045(09)70329-8. Epub 2009 Nov 10. PMID 19910250
- [Background] IJspeert JE, Bastiaansen BA, van Leerdam ME, Meijer GA, van Eeden S, Sanduleanu S, Schoon EJ, Bisseling TM, Spaander MC, van Lelyveld N, Bargeman M, Wang J, Dekker E; Dutch Workgroup serrAted polypS & Polyposis (WASP). Development and validation of the WASP classification system for optical diagnosis of adenomas, hyperplastic polyps and sessile serrated adenomas/polyps. Gut. 2016 Jun;65(6):963-70. doi: 10.1136/gutjnl-2014-308411. Epub 2015 Mar 9. PMID 25753029
- [Background] Hewett DG, Kaltenbach T, Sano Y, Tanaka S, Saunders BP, Ponchon T, Soetikno R, Rex DK. Validation of a simple classification system for endoscopic diagnosis of small colorectal polyps using narrow-band imaging. Gastroenterology. 2012 Sep;143(3):599-607.e1. doi: 10.1053/j.gastro.2012.05.006. Epub 2012 May 15. PMID 22609383
- [Derived] Bae JH, Lee C, Kang HY, Kwak MS, Doo EY, Seo JY, Song JH, Yang SY, Yang JI, Lim SH, Yim JY, Lim JH, Chung GE, Chung SJ, Jin EH, Park B, Kim JS. Improved Real-Time Optical Diagnosis of Colorectal Polyps Following a Comprehensive Training Program. Clin Gastroenterol Hepatol. 2019 Nov;17(12):2479-2488.e4. doi: 10.1016/j.cgh.2019.02.019. Epub 2019 Feb 14. PMID 30772588
- [Derived] Vleugels JLA, Dijkgraaf MGW, Hazewinkel Y, Wanders LK, Fockens P, Dekker E; DISCOUNT study group. Effects of Training and Feedback on Accuracy of Predicting Rectosigmoid Neoplastic Lesions and Selection of Surveillance Intervals by Endoscopists Performing Optical Diagnosis of Diminutive Polyps. Gastroenterology. 2018 May;154(6):1682-1693.e1. doi: 10.1053/j.gastro.2018.01.063. Epub 2018 Feb 6. PMID 29425923